CLINICAL TRIAL: NCT03974711
Title: Rampart Duo Clinical (RaDical) Study: An Exempt Minimal Risk Post-Market Evaluation of Clinical Outcomes
Brief Title: Rampart Duo Clinical (RaDical) Post-Market Study
Acronym: RaDical
Status: Completed | Type: Observational
Sponsor: Spineology, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 62-229
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All study subjects: Note: No interventions are administered under this evaluation.
  This is a real-world population. The determination to undergo a lateral lumbar interbody fusion procedure is made outside of this evaluation and is a standard of care, on-label procedure.
  Interventions: Other: In this evaluation, no interventions are performed. It is a data collection effort only. The "procedure" for this study is the data collection effort.

INTERVENTIONS:
Other: In this evaluation, no interventions are performed. It is a data collection effort only. The "procedure" for this study is the data collection effort. — There is no intervention performed in this evaluation. Data is being collected in an on-label standard of care lateral lumbar interbody fusion procedure.

SUMMARY:
This exempt, minimal risk, prospective, post-market, registry, multi-center, Institution Review Board (IRB) approved observational clinical evaluation was conducted at 10 centers. A total of 197 patients were enrolled. The evaluation collected data in a real-world patient population and was a data collection initiative only. No patient treatments or care were performed as a component of the protocol. All patient care received was on-label and standard of care for lateral lumbar interbody fusions. The data collected in this evaluation is intended to contribute to the body of literature for lateral lumbar interbody fusions.

DETAILED DESCRIPTION:
The purpose of this study was to collect data that reports on the clinical outcomes of patients that were treated with the Spineology Rampart DUO device in a standard of care instrumented lateral lumbar interbody fusion procedure at one or two contiguous levels from L2-L5. Data was collected prospectively at specified time points per protocol and included both objective and subjective measures. The study concluded when the final patient achieved their 12-month evaluation.

ELIGIBILITY:
Inclusion Criteria:

* A clinical decision has been made to treat the patient with the Rampart Duo Interbody Spacer prior to enrollment into this research evaluation. This decision is independent (made outside) of the decision to take part in the research.

Exclusion Criteria:

* Previous interbody fusion or total disc replacement at the index level(s).
* Enrolled in a concurrent clinical investigation that may confound the findings of the present investigation.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world population consistent with cleared labeling for the product.
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Short-term objective 1: New onset of thigh symptoms -- Anterior Thigh Pain Change from Baseline | 3 months
  Change from Baseline anterior thigh pain score through 3-months. Pain assessment captured on 100 mm VAS. A higher VAS score represents a worsening of pain.
Short-term objective 1: New onset of thigh symptoms -- Thigh Neurological Change from Baseline | 3 months
  Change from baseline in anterior thigh neurological assessment through 3 months. Anterior Thigh Neurological deficit defined as a negative change in strength (hip/flexor weakness) or sensation (anterior thigh).
Short-term objective 2: Hospital economics -- Blood Loss | EBL collected at time of surgery.
  Estimated blood loss (EBL) shall be compared to published literature.
Short-term objective 2: Hospital economics -- Duration of Surgery | DoS collected at time of surgery.
  Duration of surgery (DoS) defined as time from incision to closure shall be compared to published literature.
Short-term objective 2: Hospital economics -- Time-to-Discharge | Perioperative.
  Time-to-discharge (TTD) defined as time from hospital admission to the time the subject is discharged from the hospital and it shall be compared to published literature.
Long-term objective 1: Patient Low back pain change over time | Through 12 months postoperative.
  Pain measured on 100 mm VAS and compared to baseline.
Long-term objective 1: Patient Low back function change over time | Through 12 months postoperative.
  Low back function determined on Oswestry Disability Index (ODI) and compared to baseline.

SECONDARY OUTCOMES:
Additional Outcomes 1 - Radiographic Assessments | Assessed at 12 months postoperative.
  Assess for fusion status

CONTACTS AND LOCATIONS:
Overall Officials: Donald Erickson, MD, Study Chair — Retired
Locations (10):
- United States (10):
  - Bell Neuroscience Institute/Washington Township Medical Foundation, Fremont, California
  - Loma Linda University, Loma Linda, California
  - Napa Valley Orthopaedic Medical Group, Napa, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - South Florida Spine & Orthopedics, Coconut Creek, Florida
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Orthopedic Institute of Pennsylvania, Camp Hill, Pennsylvania
  - Austin Spine Specialists, Austin, Texas
  - Spine Works Institute, North Richland Hills, Texas

IPD SHARING:
Plan to Share IPD: No
IPD will be shared with study researchers for purposes of publication and presentation purposes.